CLINICAL TRIAL: NCT04548661
Title: CLinical Evaluation of Adults UNdergoing Elective Surgery Utilizing Intraoperative Incisional Wound Irrigation: A Randomized Controlled Trial (CLEAN Wound)
Brief Title: Clinical Evaluation of Adults Undergoing Elective Surgery Utilizing Intraoperative Incisional Wound Irrigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Paul Karanicolas, Scientist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CTO Project ID 4304
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Surgical Site Infection
Keywords: Intraoperative incisional wound irrigation
MeSH Terms: conditions — Surgical Wound Infection | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Pragmatic, multicentre, participant and adjudicator-blinded, three-arm randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Povidone-iodine solution (Experimental)
  Interventions: Procedure: Intraoperative incisional wound irrigation with povidone-iodine solution
- Saline (Placebo Comparator)
  Interventions: Procedure: Intraoperative incisional wound irrigation with saline
- No irrigation (No Intervention): Standard incision management

INTERVENTIONS:
Procedure: Intraoperative incisional wound irrigation with povidone-iodine solution — Participants randomized to the povidone-iodine irrigation group will have all incisions irrigated once with povidone-iodine diluted in 0.9% sterile normal saline (to a final concentration of 5% povidone-iodine (0.5% available iodine)) delivered through a bulb syringe. The povidone-iodine irrigation should be left on for 60 seconds and then dried with sterile gauze. Irrigation will be performed after any/all deep tissue layers are closed, prior to skin closure. The volume used will be left to the discretion of the clinician and irrigation will be administered until saturation is achieved.
  Arms: Povidone-iodine solution
Procedure: Intraoperative incisional wound irrigation with saline — Participants randomized to the saline irrigation group will have all incisions irrigated once with 0.9% sterile normal saline delivered through a bulb syringe. Irrigation will be performed after any/all deep tissue layers are closed, prior to skin closure. The volume used will be left to the discretion of the clinician and irrigation will be administered until saturation is achieved.
  Arms: Saline

SUMMARY:
A surgical site infection (SSI) is an infection that occurs after a surgical procedure. Despite a variety of infection prevention strategies, SSIs still occur often and impose a significant burden on patients and the healthcare system. Intraoperative irrigation (or washing of the surgical incision before closure) may reduce SSIs, but this is uncertain.

The Clinical Evaluation of Adults Undergoing Elective Surgery Utilizing Intraoperative Incisional Wound Irrigation (CLEAN Wound) trial aims to determine if incisional wound irrigation with an antiseptic or salt water solution can reduce SSIs within 30 days of surgery compared to no wound irrigation. 2,500 patients aged 18 years or older who are planned to undergo an abdominal or groin open or laparoscopic procedure will be randomly assigned to incisional wound irrigation with povidone-iodine solution; or incisional wound irrigation with saline; or no irrigation and followed for 30 days after surgery to assess the incidence of SSIs, with additional outcomes collected up to 90 days after surgery.

Even with significant advances in medicine over the past decades, there are still many fundamental issues in perioperative care that remain unclear due to lack of evidence. If this trial were to demonstrate that intraoperative wound irrigation reduces the incidence of SSI, these practice-changing findings could greatly benefit patients worldwide.

DETAILED DESCRIPTION:
Background/Rationale: Recent international guidelines and reviews have highlighted that studies of intraoperative irrigation were conducted in small samples over 30 years ago and no longer reflect the standard of care, judging the evidence to be of very low to moderate quality, and have called for additional RCTs. For example, as per the WHO Guidelines, RCTs are needed to assess frequently utilized irrigation solutions and their effect on SSI risk and state that a suitable alternative to povidone-iodine is currently unknown. Furthermore, determining whether irrigation with antiseptics and antibiotics can reduce SSIs was listed as a key research recommendation by NICE, in addition to determining cost-effectiveness of the intervention. Additional evidence is therefore required to support or refute the effectiveness of intraoperative irrigation in reducing SSIs and to address practice heterogeneity, with a focus on establishing whether irrigation is needed, and if so, which solution should be used.

Objectives: The primary objective is to determine if intraoperative incisional wound irrigation with povidone-iodine or saline in participants undergoing surgery can reduce incisional SSIs within 30 days of surgery compared to no irrigation. The secondary outcomes include: quality of life (QoL), proportion of participants prescribed systemic antibiotics, wound care received via home care services (all within 30 days of surgery); length of stay (LOS) during index hospitalization; wound dehiscence requiring reoperation, postoperative complications, mortality and healthcare utilization (all within 90 days of surgery), including: number of re-interventions (i.e. radiologically guided drain insertion or revision); number of all-cause reoperations; number of all-cause emergency department visits; number of all-cause family physician or walk-in clinic visits; and number of all-cause readmissions and length of stay of each readmission.

Study Design: This is a multicentre, pragmatic, participant and adjudicator-blinded, three-arm RCT. Participants will be randomized using an adaptive design to incisional wound irrigation with povidone-iodine versus incisional wound irrigation with saline versus no irrigation and will be followed until 30 days after surgery to assess the incidence of SSIs, with additional outcomes collected up to 90 days after surgery. The trial is adaptive, in that one of the arms may be discontinued as the trial progresses if it reaches a threshold for inferiority, and will be a continuation of our pilot trial (i.e., a vanguard design).

ELIGIBILITY:
All participants must meet all of the following inclusion criteria to participate in this study:

1. Aged 18 years or older;
2. Ontario Health Insurance Plan (OHIP) holder (for Ontario sites)

   And planned to undergo any one of the following surgical procedures:
3. a) Laparotomy, CDC Class II (clean-contaminated) or III (contaminated) incision b) Laparoscopy with a planned extraction site ≥3 cm, CDC Class II (clean-contaminated) or III (contaminated) incision c) Groin incision for open or hybrid arterial procedure

All participants meeting any of the following exclusion criteria at baseline will be excluded from participation in this study:

1. Contraindication to receiving povidone-iodine irrigation (i.e., known allergy)
2. Any active skin or soft tissue infection (at any site, including gangrene)
3. Known or anticipated CDC Class IV (Dirty) incision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2701 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of incisional surgical site infection (SSI) | Within 30 days of surgery
  SSI will be captured through blinded central review of postoperative healthcare records and participants' self-report (using a patient-reported outcome measure, or PROM). Participants will be considered to have a SSI if they meet either the health record review criteria (if any of the following occurred: 1) wound was opened and packed; 2) wound-specific treatment with antibiotics; or 3) a diagnosis of SSI explicitly recorded in medical record by treating clinician) OR PROM criteria [(i.e., if participant answers "Yes" to questions 2, 3 or 4: Have your surgical incision(s) been opened and packed (with gauze or bandages inside the wound) by a physician, physician assistant, nurse or nurse practitioner?; Have you been prescribed antibiotics for a problem with your surgical incision(s)?; Have you been told that your surgical incision(s) are infected by a physician, physician assistant, nurse or nurse practitioner?)]

SECONDARY OUTCOMES:
EQ-5D-5L Quality of life | within 30 days of surgery
  The EQ-5D-5L (not an abbreviation) is a widely used generic measure of health status consisting of two parts. The first part (the descriptive system) assesses health in five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each of which has five levels of response (no problems, slight problems, moderate problems, severe problems, extreme problems/unable to). The patient is asked to indicate their health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The second part of the questionnaire consists of a visual analogue scale (VAS) on which the patient rates their perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).
Proportion of participants requiring wound care (received via home care services) | within 30 days of surgery
Proportion of participants prescribed systemic antibiotics | within 30 days of surgery
Length of stay (LOS) (in days) | during hospitalization (up to day 30)
Proportion of participants with wound dehiscence requiring reoperation | within 90 days of surgery
Proportion of participants with postoperative complications | within 90 days of surgery
Mortality | within 90 days of surgery
Healthcare utilization | within 90 days of surgery
  1. Number of re-interventions (i.e. radiologically guided drain insertion or revision);
  2. Number of all-cause reoperations;
  3. Number of all-cause emergency department visits;
  4. Number of all-cause family physician or walk-in clinic visits; and
  5. Number of all-cause readmissions and length of stay of each readmission.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Karanicolas, MD PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (13):
- Canada (13):
  - Shared Health Manitoba, Winnipeg, Manitoba
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Health Sciences North, Greater Sudbury, Ontario
  - Hamilton Health Sciences - Juravinski Hospital, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - North York General Hospital, North York, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Mackenzie Health, Richmond Hill, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roke R, Lillie E, Daneman N, Mason SA, Tomlinson G, Jiang Y, Shiroky J, Puran S, Smith DE, Abou Khalil J, Kayssi A, Serrano PE, Pinchuk B, Apte SS, Lamb T, Ma G, Vogt K, Leslie K, Mutabdzic D, Gomez D, Ladha KS, Tsang M, Bennett S, Ullah SM, Holland J, Delisle M, Smith AJ, Calderone M, Herriott J, Voltan E, Sloan B, Muaddi H, Fergusson DA, Mazer CD, Kennedy E, Marshall JC, Aarts MA, Nathens AB, Karanicolas PJ. Clinical evaluation of adults undergoing elective surgery utilizing intraoperative incisional wound irrigation (CLEAN Wound): protocol for a randomised controlled trial. BMJ Open. 2025 Jul 17;15(7):e104375. doi: 10.1136/bmjopen-2025-104375. PMID 40675632